CLINICAL TRIAL: NCT06591624
Title: The Incidence and Analysis of Factors Related to Prolonged Mechanical Ventilation in Neurosurgical Patients: a Retrospective Cohort Study
Brief Title: Prolonged Mechanical Ventilation in Neurosurgical Patients:
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Associate professor, Chiang Mai University
Other Study IDs: ANE-2565-09317; Chiang Mai University (Other: Chiang Mai University)
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurosurgical Procedures; Neurosurgical Patients; Prolonged Mechanical Ventilation
Keywords: ventilator dependent; neurosurgical patient; prolonged mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- elective adult neurosurgical patients succesfully extubation after neurosurgery: succesfully extubation after neurosurgery
  Interventions: Other: remain intubation after surgery
- elective adult neurosurgical patients prolonged mechanical ventilation: prolonged mechanical ventilation
  Interventions: Other: Prolonged Mechanical Ventilation

INTERVENTIONS:
Other: Prolonged Mechanical Ventilation — The neurosurgical patients who could extubated within 24 h after surgery
  Groups: elective adult neurosurgical patients prolonged mechanical ventilation
Other: remain intubation after surgery — could not extubated after surgery and prolong mechanical ventilation for 48 hours
  Groups: elective adult neurosurgical patients succesfully extubation after neurosurgery

SUMMARY:
The study was carried out at the neurosurgical operating theater and neurosurgical intensive care unit, Maharaj Nakorn Chiang Mai University-Hospital. The study design was a retrospective Cohort study, recruited elective adult neurosurgical patients during December 1, 2021 to December 31, 2022. The patients were excluded if they had pre-operative definite airway control. The primary outcome was extubation success in the operating theater. Prolonged mechanical ventilation (PMV) means the patients who could not undergo the weaning protocol and extubation in 48 hours of surgery. The secondary outcome was the features associated with the prolonged mechanical ventilation.

DETAILED DESCRIPTION:
Extubation in operating theater after elective intracranial surgery is superlative. Early extubation strategy should be planned in preoperative period jointly with neurosurgical team. Any deviations from the plan should be identified, whether they originated from surgical aspects or anesthetic managements. The time-point for extubation in neurosurgical patients is more challenging compared to other non-brain surgeries. We identified some potential prognostic impacts to prolonged mechanical ventilation in elective neurosurgical patients.

The study was approved by the Institution Research Ethics Committee Panel 5, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand. (ANE-2565-09317). The study was carried out at the neurosurgical operating theater and neurosurgical intensive care unit, Maharaj Nakorn Chiang Mai University-Hospital. The study design was a retrospective Cohort study, recruited elective adult neurosurgical patients during December 1, 2021 to December 31, 2022. The patients were excluded if they had pre-operative definite airway control. The primary outcome was extubation success in the operating theater. Prolonged mechanical ventilation (PMV) means the patients who could not undergo the weaning protocol and extubation in 48 hours of surgery. The secondary outcome was the features associated with the prolonged mechanical ventilation. For continuous data, we used the student's t-test. For categorical data, we used the Fisher's exact or Chi-square test. Univariate analysis and multiple logistic regression were used to identified the prognostic factors. P values < 0.05 indicated statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* adult neurosurgical patients
* undergo elective surgery

Exclusion Criteria:

* already intubation before neurosurgical procedures
* tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was carried out at the neurosurgical operating theater and neurosurgical intensive care unit, Maharaj Nakorn Chiang Mai University-Hospital. The study design was a retrospective Cohort study, recruited elective adult neurosurgical patients during December 1, 2021 to December 31, 2022. The patients were excluded if they had pre-operative definite airway control such as intubation or tracheostomy.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
to be able to extubate after neurosurgery | within 24 hours after surgery
  successful extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Chiang Mai University, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No